CLINICAL TRIAL: NCT03161782
Title: The Efficacy of Proprioceptive Neuromuscular Facilitation Stretching and Static Stretching on Range of Motion, Pain and Function in Elbow Limitation
Brief Title: The Efficacy of Different Types of Stretching on Range of Motion, Pain and Function in Elbow Limitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Research Assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 910801
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Postoperative Pain; Elbow Fracture; Stiffness of Elbow, Not Elsewhere Classified
Keywords: pain; exercise; proprioceptive neuromuscular facilitation stretching; static stretching
MeSH Terms: conditions — Pain, Postoperative; Elbow Fractures; Pain; Motor Activity | interventions — Muscle Stretching Exercises; Exercise; Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Stretching group (Experimental): Each subject in PNF Stretching group will receive a treatment protocol consisting of PNF stretching, cold therapy and exercise.
  Interventions: Other: PNF stretching; Other: Exercise; Other: Cold Therapy
- Static Stretching group (Experimental): Each subject in Static Stretching group will receive a treatment protocol consisting of static stretching, cold therapy and exercise.
  Interventions: Other: Static Stretching; Other: Exercise; Other: Cold Therapy

INTERVENTIONS:
Other: PNF stretching — For hold-relax stretching, each subject in PNF Stretching group will be comfortably positioned in a supine lying position, and patient will move the joint to the end of the passive or pain-free ROM. The therapist will ask for an isometric contraction of the restricting muscle or pattern (antagonists) with emphasis on rotation. The patients will be asked to perform submaximal isometric contractions of the target muscle for 10 seconds. After the contraction, the patients will be instructed to relax for 5 seconds. The joint will be repositioned actively to the new limit of range, and then therapist will passively control the new ROM. The procedure will be repeated 10 times with 10 seconds of rest between two successive trials. Patients will be treated 2 times per week for 6 weeks.
  Arms: PNF Stretching group
Other: Static Stretching — For static stretching, each subject in Static Stretching group will be comfortably positioned in a supine lying position, and the stretching of target muscle will be maintained for 20 seconds followed by 10 seconds of rest. The procedure will be repeated 10 times with 10 seconds of rest between two successive trials. Patients will be treated 2 times per week for 6 weeks.
  Arms: Static Stretching group
Other: Exercise — Shoulder, elbow and wrist AROM exercises. Elbow flexion and extansion self-stretching exercises Elbow and wrist strengthening exercises Proprioception exercises for elbow. Grip strengthening exercises.
Other: Cold Therapy — Cold therapy will be applied over the elbow for 15 minutes in the form of cold pack after stretching and exercise protocol.

SUMMARY:
The aim of the study is to compare the efficacy of Proprioceptive Neuromuscular Facilitation (PNF) stretching and static stretching on range of motion (ROM), pain and function in elbow limitation.

DETAILED DESCRIPTION:
To compare the efficacy of PNF stretching and static stretching on ROM, pain and function in elbow limitation, forty voluntary patients with elbow limitation, aged between 18-55 years will be randomly divided into two groups: PNF Stretching group and Static Stretching group. PNF stretching will be combined with exercise and cold application in PNF Stretching group, static stretching will be combined with exercise and cold application in Static Stretching group, will be applied for 12 sessions. The patients will be assessed before and after six-week treatment. The pain on activity, at rest and at night will be assessed with Visual Analog Scale (VAS). ROM will be assesed with universal goniometer. The functional status will be evaluated by Disabilities Arm, Shoulder and Hand (DASH). Kinesiophobia and quality of life will be assessed with Tampa Scale for Kinesiophobia and Short Form-12, respectively. The Global Rating of Change will be used to evaluate patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Subjectswill be included with

* Aged between 18 and 65 years
* Elbow fracture in the six months before the study
* Elbow limitation in flexion or extension
* Being volunteer to participate
* Fractures should be managed with conservatively or surgically

Exclusion Criteria:

* Malunion or Nonunion Fracture
* Occurrence of complex regional pain syndrome, peripheric nerve injury, heterotopic ossification, myositis ossification or post-traumatic ankylosing
* Non-healing wound or infection
* Previously received physiotherapy for elbow limitation
* Having any cardiovascular diseases, neurological disorders, rheumatic diseases or psychiatric diseases
* Could not adjust to treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Functional Status | After the six-week intervention
  The functional status of the patients will be evaluated by The Disabilities of the Arm, Shoulder and Hand (DASH).

SECONDARY OUTCOMES:
Active Range of Motion (AROM) Assessment | Baseline
  The elbow's and forearm's AROM, including flexion, extansion, supination, pronation will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a universal goniometer. The process will be repeated three times in each direction, with the the average value recorded.
Active Range of Motion (AROM) Assessment | After the six-week intervention
  The elbow's and forearm's AROM, including flexion, extansion, supination, pronation will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a universal goniometer. The process will be repeated three times in each direction, with the the average value recorded.
Active Range of Motion (AROM) Assessment | 1-month follow up
  The elbow's and forearm's AROM, including flexion, extansion, supination, pronation will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a universal goniometer. The process will be repeated three times in each direction, with the the average value recorded.
Functional Status | Baseline
  The functional status of the patients will be evaluated by The Disabilities of the Arm, Shoulder and Hand (DASH).
Functional Status | 1-month follow up
  The functional status of the patients will be evaluated by The Disabilities of the Arm, Shoulder and Hand (DASH).
Pain Intensity | Baseline
  Pain intensity of the patients at rest, during activity, and at night will be assessed by Visual Analog Scale.
Pain Intensity | After the six-week intervention
  Pain intensity of the patients at rest, during activity, and at night will be assessed by Visual Analog Scale.
Pain Intensity | 1-month follow up
  Pain intensity of the patients at rest, during activity, and at night will be assessed by Visual Analog Scale.

OTHER OUTCOMES:
Quality of Life | Baseline
  Quality of life of the patients will be assessed by Short Form-12.
Quality of Life | After the six-week intervention
  Quality of life of the patients will be assessed by Short Form-12.
Quality of Life | 1-month follow up
  Quality of life of the patients will be assessed by Short Form-12.
Fear of movement (kinesiophobia) | Baseline
  Kinesiophobia of the patients will be assessed by Tampa Kinesiophobia Scale.
Fear of movement (kinesiophobia) | After the six-week intervention
  Kinesiophobia of the patients will be assessed by Tampa Kinesiophobia Scale.
Fear of movement (kinesiophobia) | 1-month follow up
  Kinesiophobia of the patients will be assessed by Tampa Kinesiophobia Scale.
Patient Satisfaction | After the six-week intervention
  Patient Satisfaction will be assessed with Global Rating of Change Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, MSc, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No